CLINICAL TRIAL: NCT00948415
Title: Evaluation of the Shape Up Rhode Island Campaign Study 5: Does Adding Behavioral Weight Control Information to Shape-Up Rhode Island Improve Outcomes?
Brief Title: Evaluation of the Shape Up Rhode Island Campaign Study 5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Professor, The Miriam Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2097-07 Study 5
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Internet
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SURI Enhanced (Experimental)
  Interventions: Behavioral: Evaluation of the Shape Up RI Campaign
- SURI Standard (Active Comparator)
  Interventions: Behavioral: Evaluation of the Shape Up RI Campaign

INTERVENTIONS:
Behavioral: Evaluation of the Shape Up RI Campaign — The SURI enhanced group will receive the standard Shape Up RI program. In addition, participants will be asked to record and report their daily calorie intake, body weight, minutes of physical activity, and pedometer steps. Participants will receive automated feedback on progress as well as a behavioral lesson delivered online during each week of the program. Participants assigned to the SURI Standard arm will receive the standard Shape Up RI program. The intervention will take place during the 12-week Shape Up RI campaign.

SUMMARY:
Obesity is a major health problem that has reached epidemic levels. Efforts are needed to develop cost-effective public health approaches for weight loss and maintenance. One such approach is to develop team-based programs that may motivate people to lose weight and/or increase their physical activity. One such program is entitled Shape-up Rhode Island (SURI). The current trial is investigating whether adding both a behavioral intervention delivered online PLUS automated feedback to self-monitoring would enhance the outcomes of SURI participants.

DETAILED DESCRIPTION:
Background: Given the epidemic of obesity, approaches to weight loss that can be applied on a community, state, or national level are needed. This project is an ongoing evaluation of Shape Up Rhode Island (SURI) program, a state-wide Internet based program involving team-based competition to increase physical activity and achieve weight loss.

Aim: To enhance the effectiveness of SURI utilizing a minimal contact intervention delivered online.

Design: SURI 2009 participants were invited to join a research study focusing on weight loss. Interested participants were randomized to two groups including a SURI Enhanced group (behavioral intervention presented in 12 weekly online presentations, daily self-monitoring, and weekly automated feedback) or a SURI Standard group (group given a list of previously existing online resources to aid with weight loss).

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Current participant in the Shape Up RI program weight loss competition

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Weight loss at the end of Shape Up RI | 3 Months

SECONDARY OUTCOMES:
Weight loss maintenance 6 months after program completion | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States